CLINICAL TRIAL: NCT05905965
Title: Efficacy of Double vs Standard Empapagliflozin Dose for METabolic syndromE tReatment (DEMETER - SIRIO 11) Study
Brief Title: Efficacy of Double vs Standard Empapagliflozin Dose for METabolic syndromE tReatment
Acronym: DEMETER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Kubica, Prof. dr hab., Collegium Medicum w Bydgoszczy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEMETER
Record Dates: First submitted 2023-05-12; First posted 2023-06-15 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; empagliflozin; adherence
MeSH Terms: conditions — Metabolic Syndrome | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin 20 mg (Experimental): Patients receiving empagliflozin 20 mg daily
  Interventions: Drug: Empagliflozin 20 mg
- Empagliflozin 10 mg (Active Comparator): Patients receiving empagliflozin 10 mg daily
  Interventions: Drug: Empagliflozin 10 mg

INTERVENTIONS:
Drug: Empagliflozin 20 mg — Patients receiving empagliflozin 20 mg daily - experimental arm
  Arms: Empagliflozin 20 mg
Drug: Empagliflozin 10 mg — Patients receiving empagliflozin 10 mg daily - control arm
  Arms: Empagliflozin 10 mg

SUMMARY:
The DEMETER - SIRIO 11 study is a phase III, multicenter, randomized, open-labled, investigator-initiated clinical trial with a 6 month follow-up.

The study population will include 200 subjects with diagnosis of metabolic syndrome.

All enrolled patients (nn=200) will be randomly assigned in 1:1 ratio to one of the two study arms:

1. Empagliflozin 20 mg - experimental arm
2. Empagliflozin 10 mg - control arm. Primary co-endpoints of the study include: BMI and HbA1c. Secondary endpoints include: LDL-C, triglycerides, CRP, NT-proBNP, LVEF (echocardiography), body composition, VO2max (ergospirometry), waist-hip ratio (WHR), liver steatosis assessment (LSA) by computed tomography (CT), major adverse cardiovascular events - MACE (based on medical history: heart attack, stroke, death), cardiovascular hospitalizations.

DETAILED DESCRIPTION:
The DEMETER - SIRIO 11 study is a phase III, multicenter, randomized, open-labled, investigator-initiated clinical trial with a 6 month follow-up.

The study population will include 200 subjects with diagnosis of metabolic syndrome.

All enrolled patients (nn=200) will be randomly assigned in 1:1 ratio to one of the two study arms:

1. Empagliflozin 20 mg - experimental arm
2. Empagliflozin 10 mg - control arm.

Primary co-endpoints of the study include: BMI and HbA1c.

Secondary endpoints include:

* LDL-C,
* triglycerides,
* CRP,
* NT-proBNP,
* LVEF (echocardiography),
* body composition,
* VO2max (ergospirometry),
* waist-hip ratio (WHR),
* liver steatosis assessment (LSA) by computed tomography (CT),
* major adverse cardiovascular events - MACE (based on medical history: heart attack, stroke, death),
* cardiovascular hospitalizations.

Other variables that are scheduled to be analyzed: central arterial pressure, pulse wave propagation speed, ABPM (ambulatory blood pressure monitoring), endothelial function assessment by Endopath, autonomic nervous system assessment (ANSA) by Task Force Touch CARDIO (TFTC), exercise tolerance, thickness of the adipose tissue (skin fold), blood samples: blood count, serum creatinine and eGFR, ALT, AST, GGTP, total cholesterol, HDL-C, uric acid, plasma concentration of calcium, phosphate, parathormon, 25-OH-D3, cystatin C, erythropoietin; morning urine: N-acetyl-beta-D-glucosaminidase, sodium/creatinine ratio, calcium/creatinine ratio, albumin/creatinine ratio. Moreover, functioning in chronic disease and adherence to medication and diet will be assessed with dedicated questionairies (FCIS, ACDS, ACDS diet).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of metabolic syndrome as follows: the presence of obesity (waist circumference ≥ 88 cm in women; ≥102 cm or body mass index (BMI) ≥30 kg/m2) and two of the three following criteria:

  1. high blood pressure (systolic blood pressure - in-office measurement: ≥ 130 and/or diastolic blood pressure ≥85 mm Hg or systolic blood pressure - ambulatory measurement: ≥130 and/or diastolic blood pressure ≥ 80 mm Hg) or on anti-hypertensive treatment;
  2. impaired glucose metabolism (fasting glucose ≥100 mg/dL or ≥ 140 mg/dL after 120 min in oral glucose tolerance test or HbA1c ≥5.7%) or on glucose-lowering drug treatment;
  3. elevated non-high-density lipoprotein (non-HDL ≥130 mg/dL) cholesterol level (atherogenic dyslipidemia) or on lipid-lowering drug treatment

Exclusion Criteria:

* current treatment with SGLT2 inhibitor
* chronic kidney disease with estimated glomerular filtration rate (eGFR) < 30 mL/min or on dialysis
* severely impaired liver function
* known hypersensitivity to the active empagliflozin or to any of the excipients contained in Jardiance
* history of ketoacidosis
* diabetes treated with insulin
* pregnancy
* decompensated heart failure
* acute coronary syndrome
* active thromboembolic disease
* current treatment for neoplastic disease
* active inflammatory disease within 1 month prior to enrollment
* expected lifetime <1 year
* non-cooperative patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
BMI (Body Mass Index) | 0-6 months
  change in BMI between study arms
concentration of HbA1c (glycated hemoglobin) | 0-6 months
  change in glycated hemoglobin plasma concentration between study arms

SECONDARY OUTCOMES:
concentration of LDL-C (low density cholesterol serum concentration) | 0-6 months
  change in low density cholesterol serum concentration between study arms
concentration of triglycerides | 0-6 months
  change in triglycerides serum concentration between study arms
concentration of CRP (c-reactive protein) | 0-6 months
  change in CRP serum concentration between study arms
concentration of NT-proBNP | 0-6 months
  change in NT-pro BNP serum concentration between study arms
LVEF - left ventricle ejection fraction (echocardiography) | 0-6 months
  change in LVEF (presented in percentage) between study arms
body composition analysis - body fat mass [kg] | 0-6 months
  evaluation of body fat mass [kg] change throughout the study
body composition analysis - body fat mass [%] | 0-6 months
  evaluation of body fat mass [%] change throughout the study
body composition analysis - lean body mass [kg] | 0-6 months
  evaluation of lean body mass [kg] change throughout the study
body composition analysis - lean body mass [%] | 0-6 months
  evaluation of lean body mass [%] change throughout the study
body composition analysis - skeletal muscle mass [kg] | 0-6 months
  evaluation of skeletal muscle mass [kg] change throughout the study
body composition analysis - total body water [liters] | 0-6 months
  evaluation of total body water [liters] change throughout the study
body composition analysis - total body water [%] | 0-6 months
  evaluation of total body water [%] change throughout the study
body composition analysis - extracellular water [liters] | 0-6 months
  evaluation of extracellular water [liters] change throughout the study
body composition analysis - extracellular water [%] | 0-6 months
  evaluation of extracellular water [%] change throughout the study
body composition analysis - hydration [%] | 0-6 months
  evaluation of hydration [%] change throughout the study
body composition analysis - visceral fat level [liters] | 0-6 months
  evaluation of visceral fat level [liters] change throughout the study
level of maximal oxygen uptake (VO2max) measured in ergospirometry | 0-6 months
  change in VO2 max between study arms
waist-hip ratio (WHR) | 0-6 months
  change in waist-hip ratio between study arms
liver steatosis assessment (LSA) by computed tomography (CT) | 0-6 months
  evaluation of liver steatosis assessment (LSA) assessed with computed tomography (CT), between study arms throughout the study
major adverse cardiovascular events - MACE | 0-6 months
  rate of MACE (based on medical history: heart attack, stroke, death) between study arms throughout the study
cardiovascular hospitalizations | 0-6 months
  rate of cardiovascular hospitalizations between study arms

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, Prof., Principal Investigator — Collegium Medicum w Bydgoszczy
Locations (1):
- Cardiology Department, Dr. A. Jurasz University Hospital, Bydgoszcz, Cuiavian-Pomeranian, Poland

IPD SHARING:
Plan to Share IPD: No